CLINICAL TRIAL: NCT03780790
Title: A Prospective Randomized Trial Comparing Analgesic Effects of Three Ultrasound-guided Regionel Anesthetic Techniques in Pediatrics: Caudal Analgesia, Transversus Abdominis Plane and Quadratus Lumborum Blocks
Brief Title: Comparing Analgesic Effects of Three Ultrasound Guided Regional Anesthetic Techniques in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associated Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2018/1076
Record Dates: First submitted 2018-11-20; First posted 2018-12-19 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia, Local
Keywords: quadratus lumborum block; transversus abdominis plane block; caudal block; ultrasound-guided
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: RANDOMISED DOUBLE BLINDED INTERVENTIONAL
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Quadratus Lumborum Block (Active Comparator): US-guided quadratus lumborum block will be performed with 0,5 ml/kg 0.25% Bupivacaine in the anterior layer of the thoracolumbar fascia between psoas major and quadratus lumborum muscles
  Interventions: Drug: Bupivacaine
- Transversus Abdominis Plane Block (Active Comparator): US- guided transversus abdominis plane block will be performed with 0,5 ml/kg 0.25% Bupivacaine into the fascial plane between internal oblique muscle and transversus abdominis muscle
  Interventions: Drug: Bupivacaine
- Caudal Block (Active Comparator): US-guided caudal epidural block will be applied to 0.7 ml/kg 0.25 % Bupivacaine up to a maximum of 20 mL
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — % 0,25
  Other Names: Marcaine

SUMMARY:
This study evaluates analgesic effects of ultrasound-guided (USG) regional anesthetic techniques; caudal block , transversus abdominis plane (TAP) block and quadratus lumborum block (QLB) by comparing postoperative pain scores [ Face, Legs, Activity, Cry, Consolabilty(FLACC) and Visual Analogue Scale (VAS)], first analgesic requirement time and total analgesic consumption in pediatrics undergoing lower abdominal surgery. We also aim to observe the side effects of these techniques such as nausea, vomiting, bradycardia, hypotension, respiratory depression.

DETAILED DESCRIPTION:
Lower abdominal surgeries affect dermatomes T10-L1 and blocking these nerve roots provides effective postoperative analgesia. Neuroaxial blocks such as epidural and caudal blocks is considered the gold standart regional technique for pain management after lower abdominal surgery, blocking both somatic and visceral pain. Nowadays,US is increasingly used to perform caudal block, demostrating cannule placement and precise deposition of local anesthetic in the epidural space. On the other side truncal blocks as US-guided TAP block covers T10-L1 dermatomes and provides postoperative pain relief after lower abdominal surgery with lower complication rate rather than caudal block but it may not prevent traction on the peritoneal sac. QLB is rather a new regional technique blocking nerve roots close to paravertebral area affecting somatic and visceral nerve fibers. In our study we aim to compare postoperative analgesic effects of these three techniques in paediatrics. Our primary outcomes are pain scores(FLACC/VAS) and first additional analgesic requirement time. Secondary outcomes are total analgesic consumption, side effects (nausea, vomiting, itching, urinary retention, bradycardia, hypotension, respiratory depression), length of hospitalization and chronic pain due to incision after 2 months.

ELIGIBILITY:
Inclusion Criteria:

* undergoing lower abdominal surgery
* ASA(American Society of Anestesiology)1-2

Exclusion Criteria:

* denial of patient or parents,
* infection on the local anesthetic application area
* infection in central nervous system
* coagulopathy
* brain tumours
* known allergy against local anesthetics
* anatomical difficulties
* with preexisting cardiac dysfunction
* with history of renal and/or hepatic dysfunction

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Face, Legs Activity, Cry, Consolability (FLACC) scores | up to 48 hours
  It includes five categories of behavior, each scored on 0-2 point scale so that total score ranges from 0 to 10. Total scores of 0-3 is defined as mild or no pain, 4-7 as moderate, and 8-10 as severe pain.

SECONDARY OUTCOMES:
Hospital stay | Through study completion, an average of 1 week
  Hospitalisation
Number of patients who require rescue analgesic | up to 48 hours
  Number of patients who require IV tramadol (1 mg/kg) at the first 2 hours and parasetamol in the 48 hours
First analgesic requirement time | Up to 48 hours
  Duration of postoperative analgesia

OTHER OUTCOMES:
Incidence of side effects | up to 48 hours
  Nausea, vomiting
Incidence of complications | up to first week
  Hematoma, dural puncture, infections
Time to first mobilization | up to 48 hours
  Time to first mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Principal Investigator — Istanbul University Faculty of Medicine Department of Anesthesiology
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Rectus sheath and transversus abdominis plane blocks in children: a systematic review and meta-analysis of randomized trials. — https://www.ncbi.nlm.nih.gov/pubmed/26846889
- See also: Comparison of caudal epidural block and ultrasonography-guided transversus abdominis plane block for pain relief in children undergoing lower abdominal surgery. — https://www.ncbi.nlm.nih.gov/pubmed/27555187
- See also: Quadratus Lumborum Block Versus Transversus Abdominis Plane Block in Children Undergoing Low Abdominal Surgery: A Randomized Controlled Trial. — https://www.ncbi.nlm.nih.gov/pubmed/28759502
- See also: Ultrasound-Guided Transversus Abdominis Plane and Quadratus Lumborum Blocks — https://www.nysora.com/ultrasound-guided-transversus-abdominis-plane-quadratus-lumborum-blocks